CLINICAL TRIAL: NCT06976359
Title: The National Health and Nutrition Examination Survey
Brief Title: Association of C-reactive Protein-albumin-lymphocyte Index (CALLY) With All-cause Mortality in Diabetic Patients
Acronym: required
Status: Completed | Type: Observational
Sponsor: Kunming Children's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Tian, clinician, Kunming Children's Hospital
Other Study IDs: 20250508CALLY; The 14th Five-Year Plan Yunnan (Other: Kunming Children's Hospital)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — HDL, TC, BUN,SCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on retrospective cohort data from 3,988 diabetic patients in the NHANES database, this study is the first to show a significant negative correlation between the CALLY index and all-cause mortality in diabetic patients, with good predictive ability for their survival risk. Our findings can help clinicians better assess disease progression in diabetic patients and provide a reference for personalized, precision medicine.

DETAILED DESCRIPTION:
All analyses accounted for NHANES sample weights, clustering, and stratification. We used EmpowerStats (v4.1, www.empowerstats.com) and R software (v4.4.1, www.r-project.org). Continuous variables were expressed as weighted mean ± standard error (SE), and categorical variables as weighted percentages. Associations between the CALLY index and all-cause mortality were assessed using Cox proportional hazards models. Model 1 was the unadjusted crude model. Model 2 included adjustments for age, sex, race, BMI, PIR, education, smoking, and alcohol consumption. Model 3 was the fully adjusted model including additional covariates, HDL, TC, BUN, uric acid, SCR, physical activity, energy intake, hypertension, CVD. Kaplan-Meier survival curves were used to compare survival across CALLY quartiles; differences were assessed using log-rank tests. Nonlinear associations were examined with smoothed curve fitting. Subgroup analyses explored consistency across strata. ROC curves and AUC were used to compare the predictive performance of CALLY, SII, PLR, and NLR. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

(1) self-reported doctor-diagnosed diabetes; (2) fasting blood glucose ≥ 7.0 mmol/L; (3) two-hour oral glucose tolerance test blood glucose ≥ 11.1 mmol/L; (4) glycated hemoglobin A1c (HbA1c) ≥ 6.5%; or (5) use of hypoglycemic medication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included 3,988 participants, with 1,821 deaths (weighted mortality rate: 41.7%) during a median follow-up of 131 months. Table 1 shows the baseline characteristics of participants, stratified by final mortality status. Compared to survivors, non-survivors were older (68.34 vs. 57.26 years), had a higher proportion of males (52.70% vs. 49.34%), lower educational attainment (38.15% vs. 24.50%), and higher rates of comorbid hypertension (69.44% vs. 60.50%) and cardiovascular disease (42.34% vs. 15.50%). Non-survivors also had a lower ln CALLY index (0.82 vs. 1.02, p = 0.0006). Other differences are shown in Table 1.
Sampling Method: Probability Sample
Enrollment: 3988 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
mortality | 2025-5-8
  all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Children's Hospital, Kunming, Yunnan, China